CLINICAL TRIAL: NCT04838444
Title: An Open-Label, Single Arm Trial To Evaluate Antibody Persistence And Long Term Safety Of A Live-Attenuated Chikungunya Virus Vaccine (VLA1553) In Adults Aged 18 Years and Above
Brief Title: Antibody Persistence And Long Term Safety Of A Chikungunya Virus Vaccine (VLA1553)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VLA1553-303
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VLA1553 (Experimental)
  Interventions: Biological: VLA1553

INTERVENTIONS:
Biological: VLA1553 — Trial participants previously vaccinated with VLA1553 in trial VLA1553-301 will be followed up for safety and immunogenicity.

SUMMARY:
In this open-label Phase 3b, single arm trial, persistence of antibodies and long term safety will be evaluated in up to 375 participants rolled over from trial VLA1553-301 (NCT number: NCT04546724).

DETAILED DESCRIPTION:
In this open-label Phase 3b, single arm trial, persistence of antibodies and long term safety in up to 375 participants rolled over from trial VLA1553-301 (NCT number: NCT04546724)

These participants will have annual follow-up visits at Months 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 after immunization. The primary objective of this trial will be to evaluate persistence of antibodies annually from 1 to 10 years after the single immunization with VLA1553. The secondary objective is to evaluate long-term safety 6 months to 2 years after the single immunization with VLA1553.

ELIGIBILITY:
Inclusion Criteria:

* Individual participated in the VLA1553-301 clinical trial;
* Participant has an understanding of the trial and its procedures, agrees to its provisions, and voluntarily gives written informed consent prior to any trial-related procedures;
* Participant had immunogenicity blood samples taken at baseline (Visit 1) and either Day 29 (Visit 3), Day 85 (Visit 4) or Day 180 (Visit 5) in Trial VLA1553-301 and was negative for neutralizing antibodies at baseline

Exclusion Criteria:

* Participant presents with clinical conditions representing a contraindication to blood draws;
* Participant has donated blood or use of blood products prior 30 days of immunogenicity sampling;
* Participant has received an active drug with potential immunosuppressive action or investigational drug or device within a period of 30 days prior a trial visit;
* Participant has a known or suspected problem with alcohol or drug abuse as determined by the Investigator;
* Participant has any condition that, in the opinion of the Investigator, may compromise the participant's well-being, might interfere with evaluation of trial endpoints, or would limit the participant's ability to complete the trial;
* Participant is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
* Participant is a member of the team conducting the trial or in a dependent relationship with one of the trial team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with seroresponse levels post-vaccination. (defined as µPRNT50 ≥150) | until Year 10

SECONDARY OUTCOMES:
Frequency of any Serious Adverse Event (SAE) | until Year 2
Relatedness of any Serious Adverse Event (SAE) | until Year 2
Immune response as measured by CHIKV-specific neutralizing antibody titers post-vaccination | until Year 10
Proportion of participants with seroconversion | until Year 10
Fold increase of CHIKV-specific neutralizing antibody titers post-vaccination as compared to baseline (i.e. at start of trial VLA1553-301) | until Year 10
Proportion of participants reaching an at least 4-fold, 8-fold, 16-fold or 64-fold increase in CHIKV-specific neutralizing antibody titer compared to baseline | until Year 10

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (10):
- United States (10):
  - Accelerated Enrollment Solutions (AES), Phoenix, Arizona
  - Velocity Clinical Research, Hallandale, Florida
  - Accelerated Enrollment Solutions (AES), Chicago, Illinois
  - Alliance for Multispecialty Research (AMR), Lexington, Kentucky
  - Velocity Clinical Research, Grand Island, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Alliance for Multispecialty Research (AMR), Knoxville, Tennessee
  - Velocity Clinical Research, Austin, Texas
  - Velocity Clinical Research, West Jordan, Utah
  - Allliance for Multispecialty Research (AMR), Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
After trial completion, Valneva may provide access to individual de-identified participant data and related trial documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Trial Report (CTR)) upon request from qualified researchers, and subject to Valneva's review and approval.

REFERENCES:
- [Derived] McMahon R, Toepfer S, Sattler N, Schneider M, Narciso-Abraham M, Hadl S, Hochreiter R, Kosulin K, Mader R, Zoihsl O, Wressnigg N, Dubischar K, Buerger V, Eder-Lingelbach S, Jaramillo JC. Antibody persistence and safety of a live-attenuated chikungunya virus vaccine up to 2 years after single-dose administration in adults in the USA: a single-arm, multicentre, phase 3b study. Lancet Infect Dis. 2024 Dec;24(12):1383-1392. doi: 10.1016/S1473-3099(24)00357-8. Epub 2024 Aug 12. PMID 39146946